CLINICAL TRIAL: NCT02621398
Title: Moving PD-1 Blockade With Pembrolizumab Into Concurrent Chemoradiation for Locally Advanced Non-Small Cell Lung Cancer
Brief Title: Pembrolizumab, Paclitaxel, Carboplatin, and Radiation Therapy in Treating Patients With Stage II-IIIB Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Salma Jabbour, MD, Professor, Radiation Oncology, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 031507; NCI-2015-01810 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20150002247 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Results first posted 2023-10-11 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Stage II Non-Small Cell Lung Cancer; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy, Conformal; Carboplatin; Radiotherapy, Intensity-Modulated; Paclitaxel; Taxes; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (paclitaxel, carboplatin, radiation, pembrolizumab) (Experimental): Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 1, 8, 15, 22, 29, and 36. Patients undergo 3D CRT or IMRT QD 5 days a week for 6 weeks. Beginning 2-6 weeks after, 2 weeks before the end, or at the start of chemotherapy and radiation therapy, patients also receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Carboplatin; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Biological: Pembrolizumab

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D-CRT or IMRT
  Other Names: 3-dimensional radiation therapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Radiation: Intensity-Modulated Radiation Therapy — Undergo 3D-CRT or IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase I trial studies the side effects, best dose, and best way to give pembrolizumab when given together with paclitaxel, carboplatin, and radiation therapy in treating patients with stage II-IIIB non-small cell lung cancer. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving pembrolizumab together with paclitaxel, carboplatin, and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess safety and toxicity of anti-programmed cell death 1 (PD-1) inhibition with pembrolizumab with concurrent chemoradiation therapy for non-operable, locally advanced non-small cell lung cancer.

SECONDARY OBJECTIVES:

I. To evaluate local control and distant metastasis-free survival, progression-free and overall survival with the addition of pembrolizumab to chemoradiotherapy.

II. To evaluate the rates of pneumonitis that may result from combination pembrolizumab and chemoradiotherapy.

TERTIARY OBJECTIVES:

I. To assess whether programmed cell death ligand 1 (PDL1) status on immunohistochemistry is predictive of response to pembrolizumab when combined with chemoradiation therapy.

II. To assess T cell (cluster of differentiation 8 positive [CD8+] T cells and CD4+ forkhead box P3 positive [FoxP3+] regulatory cells) responses at weeks 1, 3, 6 during chemoradiation therapy and before each administration of pembrolizumab for cycles 1, 2, 3.

OUTLINE: This is a dose-escalation study of pembrolizumab.

Patients receive paclitaxel intravenously (IV) over 1 hour and carboplatin IV over 30 minutes on days 1, 8, 15, 22, 29, and 36. Patients undergo 3-dimensional (3D) conformal radiation therapy (CRT) or intensity-modulated radiation therapy (IMRT) once daily (QD) 5 days a week for 6 weeks . Beginning 2-6 weeks after, 2 weeks before the end, or at the start of chemotherapy and radiation therapy , patients also receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days every 12 weeks for 1 year, every 16 weeks for 1 year, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and Health Insurance Portability and Accountability Act (HIPPA) authorization for release of personal health information
* Subjects with any kind of non-small cell lung carcinoma (NSCLC) histology documented by histology or cytology from bronchial brushing or washing, or needle aspiration of a defined lesion but not from sputum cytology alone
* Must have American Joint Committee on Cancer (AJCC) 7th edition (ed) inoperable stage II disease requiring chemoradiation therapy or stage IIIA or IIIB NSCLC based on appropriate staging studies including brain magnetic resonance imaging (MRI) or head computed tomography (CT), CT chest, and fluorodeoxyglucose (FDG) positron emission tomography (PET)/CT scan
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion; newly-obtained is defined as a specimen obtained up to 8 weeks (56 days) before initiation of treatment on day 1; subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the sponsor or may undergo fine needle aspiration
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 14 days before registration for protocol therapy
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Serum creatinine OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance rate [CrCl]) =< 1.5 X upper limit of normal (ULN) OR >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases
* Albumin >= 2.5 mg/dL
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Forced expiratory volume >= 1.0 L or >= 40% of predicted with or without bronchodilators by pulmonary function testing
* Women of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Women of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days before the first dose of trial treatment
* Has a known history of active Bacillus tuberculosis (TB)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may not participate
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti- programmed cell death 1 ligand 2 (PD-L2) agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive) or hepatitis C (HCV) (e.g., HCV ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy
* Pleural effusion that cannot be controlled despite appropriate interventions
* History of allergy or hypersensitivity to any component of the treatment
* No active second cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salma Jabbour, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (3):
- United States (3):
  - Yale Cancer Center, New Haven, Connecticut
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jabbour SK, Berman AT, Decker RH, Lin Y, Feigenberg SJ, Gettinger SN, Aggarwal C, Langer CJ, Simone CB 2nd, Bradley JD, Aisner J, Malhotra J. Phase 1 Trial of Pembrolizumab Administered Concurrently With Chemoradiotherapy for Locally Advanced Non-Small Cell Lung Cancer: A Nonrandomized Controlled Trial. JAMA Oncol. 2020 Jun 1;6(6):848-855. doi: 10.1001/jamaoncol.2019.6731. PMID 32077891

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 2-6 Weeks -Treatment Dose Level -1; Pembrolizumab 100mg: Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 1, 8, 15, 22, 29, and 36. Patients undergo 3D CRT or IMRT QD 5 days a week for 6 weeks. Beginning 2-6 weeks after, 2 weeks before the end, or at the start of chemotherapy and radiation therapy, patients also receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.
  3-Dimensional Conformal Radiation Therapy: Undergo 3D-CRT or IMRT
  Carboplatin: Given IV
  Intensity-Modulated Radiation Therapy: Undergo 3D-CRT or IMRT
  Laboratory Biomarker Analysis: Correlative studies
  Paclitaxel: Given IV
  Pembrolizumab: Given IV
  Dose Level -1 Pembrolizumab 100mg Q3 weeks
- Arm 2-6 Weeks Post Treatment After CRT-Pembrolizumab Dose Level: 1 200mg: Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 1, 8, 15, 22, 29, and 36. Patients undergo 3D CRT or IMRT QD 5 days a week for 6 weeks. Beginning 2-6 weeks after, 2 weeks before the end, or at the start of chemotherapy and radiation therapy, patients also receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.
  3-Dimensional Conformal Radiation Therapy: Undergo 3D-CRT or IMRT
  Carboplatin: Given IV
  Intensity-Modulated Radiation Therapy: Undergo 3D-CRT or IMRT
  Laboratory Biomarker Analysis: Correlative studies
  Paclitaxel: Given IV
  Pembrolizumab: Given IV
  Dose Level 1 Pembrolizumab 200mg Q3 weeks Dose Level: 1 200mg
- 2-6 WEEKS AFTERArm: 2 Weeks Before Chemoradiation (CRT) END Dose Level: 2 Pembrolizumab 100mg: 2 weeks before the end, or at the start of chemotherapy and radiation therapy
  Dose Level: 2 Pembrolizumab 100mg Q3 weeks
- Arm: 2 Weeks Before Chemoradiation (CRT) END Dose Level: 3 Pembrolizumab 200mg: 2 weeks before the end, or at the start of chemotherapy and radiation therapy
  Dose Level: 3 Pembrolizumab 200mg Q3 weeks
- Arm: At Start of CRT Dose Level: 4 Pembrolizumab 100mg CRT Pembrolizumab 200 mg: At the start of chemotherapy and radiation therapy Dose Level: 4 Pembrolizumab 100mg Q3 weeks
- Arm: At Start of CRT Dose Level: 5 Pembrolizumab 200mg: At the start of chemotherapy and radiation therapy
  Dose Level: 5 Pembrolizumab 200mg Q3 weeks
- Arm: At Start of CRT Dose Level: 5-E Pembrolizumab 200mg: At the start of chemotherapy and radiation therapy Dose Level: 5E Pembrolizumab 200mg Q3 weeks
Period: Overall Study
Arm/Group | Arm 2-6 Weeks -Treatment Dose Level -1; Pembrolizumab 100mg | Arm 2-6 Weeks Post Treatment After CRT-Pembrolizumab Dose Level: 1 200mg | 2-6 WEEKS AFTERArm: 2 Weeks Before Chemoradiation (CRT) END Dose Level: 2 Pembrolizumab 100mg | Arm: 2 Weeks Before Chemoradiation (CRT) END Dose Level: 3 Pembrolizumab 200mg | Arm: At Start of CRT Dose Level: 4 Pembrolizumab 100mg CRT Pembrolizumab 200 mg | Arm: At Start of CRT Dose Level: 5 Pembrolizumab 200mg | Arm: At Start of CRT Dose Level: 5-E Pembrolizumab 200mg
Started | 0 | 4 | 4 | 3 | 3 | 3 | 6
Completed | 0 | 4 | 4 | 3 | 3 | 3 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: no data collect for this group
Groups:
- Arm 2-6 Weeks -Treatment Dose Level -1; Pembrolizumab 100mg: Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 1, 8, 15, 22, 29, and 36. Patients undergo 3D CRT or IMRT QD 5 days a week for 6 weeks. Beginning 2-6 weeks after, 2 weeks before the end, or at the start of chemotherapy and radiation therapy, patients also receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.
  3-Dimensional Conformal Radiation Therapy: Undergo 3D-CRT or IMRT
  Carboplatin: Given IV
  Intensity-Modulated Radiation Therapy: Undergo 3D-CRT or IMRT
  Laboratory Biomarker Analysis: Correlative studies
  Paclitaxel: Given IV
  Pembrolizumab: Given IV
- Arm: 2 Weeks Before Chemoradiation (CRT) END Dose Level: 2 Pembrolizumab 100mg: 2 weeks before the end, or at the start of chemotherapy and radiation therapy
  Dose Level: 2 Pembrolizumab 100mg Q3 weeks
- Arm: At Start of CRT Dose Level: 4 Pembrolizumab 100mg: At the start of chemotherapy and radiation therapy Dose Level: 4 Pembrolizumab 100mg Q3 weeks
- Total: Total of all reporting groups
Arm/Group | Arm 2-6 Weeks -Treatment Dose Level -1; Pembrolizumab 100mg | Arm 2-6 Weeks Post Treatment After CRT-Pembrolizumab Dose Level: 1 200mg | Arm: 2 Weeks Before Chemoradiation (CRT) END Dose Level: 2 Pembrolizumab 100mg | Arm: 2 Weeks Before Chemoradiation (CRT) END Dose Level: 3 Pembrolizumab 200mg | Arm: At Start of CRT Dose Level: 4 Pembrolizumab 100mg | Arm: At Start of CRT Dose Level: 5 Pembrolizumab 200mg | Arm: At Start of CRT Dose Level: 5-E Pembrolizumab 200mg | Total
Number analyzed (Participants) | 0 | 4 | 4 | 3 | 3 | 3 | 6 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 2 | 0 | 2 | 3 | 7
  >=65 years | 0 | 4 | 4 | 1 | 3 | 1 | 3 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 0 | 3 | 0 | 1 | 3 | 10
  Male | 0 | 1 | 4 | 0 | 3 | 2 | 3 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 3
  White | 0 | 2 | 4 | 3 | 2 | 3 | 6 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 4 | 4 | 3 | 3 | 3 | 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) and Dose Limiting Toxicity (DLT) of the Combination of Pembrolizumab With Paclitaxel, Carboplatin and Radiation Therapy According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: The 3+3 algorithm design will be used to find the MTD. Safety will be evaluated by DLT, defined as grade 4 pneumonitis. Toxicities will be characterized based on seriousness, causality, toxicity grading, and action taken with regard to trial treatment.
Time Frame: Up to 30 days
Measure: Number; unit: mg
Groups:
- All Participants: All participants who received at least one dose of Pembrolizumab; either 100mg or 200 mg.
Arm/Group | All Participants
Number analyzed (Participants) | 23
mg | 200

2. Secondary Outcome: Overall Survival as Measured by the Kaplan Meier Estimation Method
Description: Overall survival is the overall longevity of the patient from time of initiation of chemoradiation to time of death.
Time Frame: Time of initiation of chemoradiation through study completion (death)
Reporting Status: Not Posted

3. Secondary Outcome: Best Overall Response According to Response Evaluation Criteria in Solid Tumors RECIST 1.1
Description: Best response on treatment was based on RECIST 1.1. Complete response (CR) is complete disappearance of all target lesions; Partial Response (PR) is at least 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as a reference baseline sum. Progressive disease(PD) is at least 20%increase in the sum of the longest diameter of target lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions or progression of non-target lesions. Stable disease is defined as any condition not meeting the above criteria.
Time Frame: Time of initiation of chemoradiation through study completion (death)
Reporting Status: Not Posted, anticipated posting 2042-10

4. Secondary Outcome: Metastasis-free Survival as Measured by the Kaplan Meier Estimation Method
Description: The length of time from the start of treatment and cancer has not spread to other parts of the body.
Time Frame: Time of initiation of chemoradiation through study completion (death)
Reporting Status: Not Posted, anticipated posting 2042-10

5. Secondary Outcome: Progression Free Survival According Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and as Measured by the Kaplan Meier Estimation Method
Description: Progression-free survival is the event without sign of any progression either locally or distantly, measured from the initiation of chemoradiation. Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) for target lesions and assessed by CT or MRI imaging: Complete response (CR) - disappearance of all target lesions; Partial response (PR) - >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) - At least a 20% increase in the sum of the longest diameter of target lesions; or Stable Disease (SD) - neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Time of initiation of chemoradiation through study completion (death)
Reporting Status: Not Posted, anticipated posting 2042-10

6. Secondary Outcome: Immune-related Response Evaluation Criteria In Solid Tumors Using Immune-Related Response (irRC).
Description: Immune-Related Complete Response (irCR): Complete disappearance of all tumor lesions for at least 4 weeks from the date of documentation of complete response.
  Immune-Related Partial Response (irPR): The sum of the products of the two largest perpendicular diameters of all index lesions is measured and captured as the SPD baseline. At each subsequent tumor assessment, the sum of the products of the two largest perpendicular diameters of all index lesions and of new measurable lesions are added together to provide the Immune Response Sum of Product Diameters (irSPD). A decrease, relative to baseline of the irSPD compared to the previous SPD baseline, of 50% or greater is considered an immune Partial Response
  Immune-Related Stable Disease (irSD): irSD is defined as the failure to meet criteria for immune complete response or immune partial response, in the absence of progressive disease
Time Frame: Time of initiation of chemoradiation through study completion (death)
Reporting Status: Not Posted, anticipated posting 2042-10

ADVERSE EVENTS:
Time Frame: Up to 30 days
Description: no data collected for this group
Groups:
- Arm 2-6 Weeks -Treatment Dose Level -1; Pembrolizumab 100mg: Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 1, 8, 15, 22, 29, and 36. Patients undergo 3D CRT or IMRT QD 5 days a week for 6 weeks. Beginning 2-6 weeks after, 2 weeks before the end, or at the start of chemotherapy and radiation therapy, patients also receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.
  3-Dimensional Conformal Radiation Therapy: Undergo 3D-CRT or IMRT
  Carboplatin: Given IV
  Intensity-Modulated Radiation Therapy: Undergo 3D-CRT or IMRT
  Laboratory Biomarker Analysis: Correlative studies
  Paclitaxel: Given IV
  Pembrolizumab: Given IV Dose Level -1; Pembrolizumab 100mg
- Arm 2-6 Weeks -Treatment Dose Level 1; Pembrolizumab 200mg: Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 1, 8, 15, 22, 29, and 36. Patients undergo 3D CRT or IMRT QD 5 days a week for 6 weeks. Beginning 2-6 weeks after, 2 weeks before the end, or at the start of chemotherapy and radiation therapy, patients also receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.
  3-Dimensional Conformal Radiation Therapy: Undergo 3D-CRT or IMRT
  Carboplatin: Given IV
  Intensity-Modulated Radiation Therapy: Undergo 3D-CRT or IMRT
  Laboratory Biomarker Analysis: Correlative studies
  Paclitaxel: Given IV
  Pembrolizumab: Given IV Dose Level 1; Pembrolizumab 200mg
- Arm: 2 Weeks Before h Chemoradiation (CRT) END Dose Level: 2 Pembrolizumab 100mg: 2 weeks before the end, or at the start of chemotherapy and radiation therapy Dose Level 2; Pembrolizumab 100mg
- Arm: 2 Weeks Before h Chemoradiation (CRT) END Dose Level: 3 Pembrolizumab 200mg: 2 weeks before the end, or at the start of chemotherapy and radiation therapy
  Dose Level 3; Pembrolizumab 200mg
- Arm: At Start of CRT Dose Level: 4 Pembrolizumab 100mg: At the start of chemotherapy and radiation therapy
  Dose Level 4; Pembrolizumab 100mg
- Arm: At Start of CRT Dose Level: 5 Pembrolizumab 200mg: At the start of chemotherapy and radiation therapy
  Dose Level 5; Pembrolizumab 200mg
- Arm: At Start of CRT Dose Level: 5E Pembrolizumab 200mg: At the start of chemotherapy and radiation therapy
  Dose Level 5-E; Pembrolizumab 200mg
Arm/Group | Arm 2-6 Weeks -Treatment Dose Level -1; Pembrolizumab 100mg | Arm 2-6 Weeks -Treatment Dose Level 1; Pembrolizumab 200mg | Arm: 2 Weeks Before h Chemoradiation (CRT) END Dose Level: 2 Pembrolizumab 100mg | Arm: 2 Weeks Before h Chemoradiation (CRT) END Dose Level: 3 Pembrolizumab 200mg | Arm: At Start of CRT Dose Level: 4 Pembrolizumab 100mg | Arm: At Start of CRT Dose Level: 5 Pembrolizumab 200mg | Arm: At Start of CRT Dose Level: 5E Pembrolizumab 200mg
All-Cause Mortality (participants affected / at risk) | 0/0 | 4/4 | 4/4 | 1/3 | 1/3 | 2/3 | 3/6
Serious Adverse Events (participants affected / at risk) | 0/0 | 2/4 | 0/4 | 0/3 | 0/3 | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 0/0 | 4/4 | 4/4 | 3/3 | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 2-6 Weeks -Treatment Dose Level -1; Pembrolizumab 100mg (N=0) | Arm 2-6 Weeks -Treatment Dose Level 1; Pembrolizumab 200mg (N=4) | Arm: 2 Weeks Before h Chemoradiation (CRT) END Dose Level: 2 Pembrolizumab 100mg (N=4) | Arm: 2 Weeks Before h Chemoradiation (CRT) END Dose Level: 3 Pembrolizumab 200mg (N=3) | Arm: At Start of CRT Dose Level: 4 Pembrolizumab 100mg (N=3) | Arm: At Start of CRT Dose Level: 5 Pembrolizumab 200mg (N=3) | Arm: At Start of CRT Dose Level: 5E Pembrolizumab 200mg (N=6)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 2-6 Weeks -Treatment Dose Level -1; Pembrolizumab 100mg (N=0) | Arm 2-6 Weeks -Treatment Dose Level 1; Pembrolizumab 200mg (N=4) | Arm: 2 Weeks Before h Chemoradiation (CRT) END Dose Level: 2 Pembrolizumab 100mg (N=4) | Arm: 2 Weeks Before h Chemoradiation (CRT) END Dose Level: 3 Pembrolizumab 200mg (N=3) | Arm: At Start of CRT Dose Level: 4 Pembrolizumab 100mg (N=3) | Arm: At Start of CRT Dose Level: 5 Pembrolizumab 200mg (N=3) | Arm: At Start of CRT Dose Level: 5E Pembrolizumab 200mg (N=6)
Respirtory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (14) | 4 (36) | 3 (9) | 3 (18) | 1 (2) | 6 (52)
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 4 (13) | 3 (33) | 3 (12) | 2 (6) | 3 (16) | 6 (33)
General disorders and administration site conditions (General disorders) | 0 (0) | 4 (9) | 2 (17) | 2 (11) | 2 (12) | 2 (15) | 6 (18)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 (0) | 3 (9) | 4 (10) | 1 (5) | 1 (3) | 3 (7) | 3 (5)
Infections and infestations (Infections and infestations) | 0 (0) | 2 (3) | 4 (10) | 1 (2) | 1 (3) | 1 (1) | 5 (7)
Nervous system disorders (Nervous system disorders) | 0 (0) | 1 (1) | 2 (10) | 2 (2) | 2 (4) | 2 (5) | 6 (10)
Investigations (Investigations) | 0 (0) | 2 (6) | 3 (16) | 1 (13) | 2 (16) | 2 (7) | 1 (4)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (4) | 2 (5) | 2 (10) | 2 (2) | 3 (3)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 1 (2) | 2 (5) | 1 (2) | 2 (3) | 3 (3)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (17) | 1 (3) | 2 (8) | 0 (0) | 2 (2)
Endocrine disorders (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 2 (6)
Renal (Renal and urinary disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vascular (Vascular disorders) | 0 (0) | 1 (3) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
Aside from the use of only one chemotherapy doublet regimen, other limitations of this study are the small sample size and limited follow-up duration. This study, although multi institutional, was performed at only three institutions. Also, participants may have received photon therapy or proton therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol: study protocol (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT02621398/Prot_000.pdf
  • Study Protocol and Statistical Analysis Plan: study protocol SAP 2 (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT02621398/Prot_SAP_001.pdf
  • Informed Consent Form (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/98/NCT02621398/ICF_002.pdf